CLINICAL TRIAL: NCT03564041
Title: Alternative Treatments to Help Late-Life Depression Study Protocol
Brief Title: SSM vs HEP in Late-Life Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4961
Record Dates: First submitted 2018-05-16; First posted 2018-06-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Late-life Depression; Treatment-resistant Depression
Keywords: depression; late-life; executive functioning; sahaj samadhi; meditation; treatment-resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Intervention Model Description: This study will be a blinded (rater, investigator, and clinician), 12-week randomized controlled trial (RCT) conducted at Western University, London, ON, Canada, and McGill University, Montreal, QC, Canada.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant enrolment will be masked from care provider, investigator, and the outcomes assessors through the use of third party randomization. This ensures that only participants, and those necessary in coordinating their participation in the study, are aware of whether or not they are part of the experimental or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sahaj Samadhi Meditation (SSM) (Experimental): SSM will be taught to participants over 4 consecutive days, for 2 hours each day. Participants will initially learn about the nature of meditation and will be taken through a guided meditation. Afterwards, participants will undergo training which includes understanding the nature of the mind and the thoughts arising from it, guided meditation by the instructor, and a discussion of what is correct and incorrect meditation. Follow-ups will be conducted once every week for the following 11 weeks, each including guided meditation. Participants will be encouraged to practice the meditation at home for 20 minutes per session and will be given weekly practice logs to complete.
  Interventions: Behavioral: Sahaj Samadhi Meditation (SSM)
- Health Enhancement Program (HEP) (Other): Arm type: Active control group
  HEP controls for several non-specific factors found in a meditation group such as Sahaj Samadhi, including: group support and morale, behavioral activation, reduction of stigma, facilitator attention, treatment duration, and time spent on at-home practice. HEP has been tailored to be structurally equivalent to a SSM intervention, with similar-sized groups, meeting for 4 days for 2 hours, and then a one-hour follow up session weekly for the subsequent 11 weeks, and completing the same amount of home practice (20 minutes twice daily, every day), and will be asked to complete weekly practice logs.
  Interventions: Behavioral: Health Enhancement Program (HEP)

INTERVENTIONS:
Behavioral: Sahaj Samadhi Meditation (SSM) — This is the experimental arm of the study, where participants will be trained in a form of meditation that may improve depressive symptoms.
  Arms: Sahaj Samadhi Meditation (SSM)
Behavioral: Health Enhancement Program (HEP) — This is the active control group of the study, where participants will be educated on health promotion, healthy diet, music, and exercise, but do not learn breathing techniques, or meditation.
  Arms: Health Enhancement Program (HEP)

SUMMARY:
The investigators will conduct a randomized controlled trial (RCT), comparing SSM (n=96) versus HEP (n=96) in 192 LLD participants stratified by site and presence of treatment resistant late life depression (TR-LLD). Participants will be blinded to the treatment hypothesis while investigators, raters and treating clinicians will be additionally blinded to the intervention. Both SSM and HEP will be taught over 4 consecutive days in similar sized groups (4-10 participants) followed by weekly reinforcement sessions for subsequent 11 weeks. Trained raters will collect data on depression symptoms (HAM-D 17 scale) and cognition at baseline, 12-week and 26-week follow-up as the primary and secondary outcome measures respectively.

DETAILED DESCRIPTION:
RECRUITMENT AND CONSENT:

Participants will either be recruited from primary-, secondary-, and tertiary-care centres or from self-referral (general public). Montreal patients will be recruited from the Douglas Institute and associated Integrated University Health and Social Services Centres (CIUSSS)-Ouest de l'ile Local Community Services Centres (CLSCs) (CLSC Verdun and CLSC Lasalle), Jewish General Hospital (JGH) Psychiatry clinics (Institute for Community and Family Psychiatry) and associated CIUSSS-Centre-Ouest family medicine clinics/CLSCs: CLSC Benny Farm, CLSC Rene Cassin, CLSC Côte Des Neiges, CLSC Metro, CLSC Parc Extension, Herzl Family Medicine JGH, St-Mary's Dept. of Psychiatry, and McGill University Health Centre (MUHC) Dept. of Psychiatry. London participants will be recruited from London Health Science Centre (LHSC) sites (Victoria Hospital and University Hospital) and Parkwood Institute - Mental Health Care Building. Participants will be screened for eligibility and given a letter of information (LOI) for their review. After 24 hours, a research assistant will contact the participant and, if they are interested in participating and eligible to participate in the research study, they will be recruited into the study after valid consent is received.

STUDY INTERVENTION:

This study is a 12-week, randomized controlled trial seeking to recruit 192 participants with late-life depression total across two sites - (1) McGill University, Montreal, Quebec (QC), and (2) University of Western Ontario in London, Ontario (ON). Participants will be randomly assigned to one of two conditions: Sahaj Samadhi Meditation (SSM) or the Health Enhancement Program (HEP). The SSM intervention will be offered by trained and certified teachers from the Art of Living Foundation at Montreal and London between August 2018 and August 2021. The HEP intervention will be offered by a trained Nurse Practitioner, Social Worker, Psychologist, Occupational Therapist or other qualified professional at Montreal and London between August 2018 and August 2022. Raters, clinicians, and care providers will be blind to participant study condition.

SSM (the experimental group) and HEP (the active control group) require participants to attend training for 4 days, attend weekly follow-up sessions, and to practice the trained techniques at home for 20-minutes per day (details of each intervention can be found below). Participants will additionally be asked to fill out "homework logs" to record days they practiced the trained technique. A total of 3 assessment sessions are planned for participants to attend: to occur at baseline (0-week) as well as at 12-week and 26-week follow-ups.

MENTAL HEALTH ASSESSMENTS:

Participants will be screened using the Screening for Cognitive Impairment in Older Adults (Mini-Cog), Patient Health Questionnaire (PHQ-9), the Magnetic Resonance Imaging (MRI) pre-screening questionnaire, the Mini International Neuropsychiatric Interview, the Test of Premorbid Functioning, and the Antidepressant Treatment History Form (ATHF). Participants will be tested for the primary outcome, depression, using the Hamilton Depression Rating Scale (HAM-D17). The secondary outcome, executive functioning, will be measured by the Wechsler Adult Intelligence Scale (WAIS) Digit Span, Delis-Kaplan (D-KEFS) Verbal Fluency Test, Rey-Osterrieth Complex Figure-Copy Trial, and the California Verbal Learning Test-II-Short Form. Measures of primary and secondary outcomes will be administered at all 3 assessment sessions. All measures are described below.

BLOOD DRAW:

Blood draws will be performed at baseline (0-weeks) and 12-week follow-up by a qualified nurse at the CLSC in Montreal and Parkwood Mental Health in London. The blood collected will be stored at the Douglas Mental Health University Institute in Montreal, QC, and at Robart's Research Institute in London, ON.

GAIT:

Gait data will be collected in London, Ontario, only. The data to be collected is weight, height, waist circumference, and hip circumference. Gait data will be measured alongside the Falls Efficacy Scale (FES-I) (described below).

MRI:

The investigators aim to recruit a total of 50 participants (25 from each group) from the SSM/HEP study into a magnetic resonance imaging (MRI) study that will involve MRI scans at baseline and at the 12-week follow-up. Participants eligible for this sub-study will have had to complete the MRI pre-screening questionnaire. Those who are part of this sub-study will be invited to attend two MRI scanning sessions, which are expected to take about 1.5 h, to occur at baseline and the 12-week follow-up. Each MRI appointment will be completed in addition to the tasks described above.

STATISTICAL ANALYSIS

Descriptive statistics will be run with continuous variables summarized using mean and standard deviations and categorical variables summarized using counts and proportions. HDRS-17 scores at baseline and 12-week follow-up of patients assigned to SSM and HEP will be compared using linear mixed models. This approach will account for the clustering of observations, since both SSM and HEP will be delivered in a group setting. Next, we will evaluate whether a greater proportion of patients assigned to SSM, compared to HEP, achieve depression remission (defined as a HDRS-17 score ≤7 at the 12-week follow-up) using generalized linear mixed models.

We will take Z-scores of executive functioning tests at baseline and at 12-week follow-up for each test and take the mean of these to calculate an overall Z-score for Planning and Organizing Cognition Measures. Z-scores at baseline and at 12-week follow-up of patients assigned to SSM and HEP will be compared using linear mixed models.

PROTOCOL DEVIATIONS

On March 22, 2019 a protocol deviation occurred when a preliminary analysis (n=14) was completed for the purpose of an undergraduate student research volunteer's course requirements. This volunteer did not have access to patient identifiers. The results were presented at an undergraduate research day as a poster with no abstract in the public domain.

This preliminary analysis has the potential to reduce the available degrees of freedom for the final study analyses. It could also be that blinded personnel (raters and PI) who are now aware of the preliminary results may inadvertently suffer from selection /outcome bias.

The investigators agree that the risk of this preliminary analysis jeopardizing the final analysis is theoretically significant and hence data from these participants will not be included in the final analyses.

On September 5, 2019 two protocol deviations occurred when all the participants in a cohort (n=4) were allocated to attend the SSM intervention. This decision was made at that time a) to maintain recruitment targets and b) to ensure the therapeutic effect of a group intervention a size of 4-6 was felt necessary.

It was felt that that if minimum group size participants are not met, participants will not benefit from the support of their peers as offered by SSM and/or HEP.

As a result of this decision two protocol violations occurred: 1. one participant did not attend the intervention to which they were randomized but rather to the other intervention 2. the study rater was unblinded to the allocations of all 4 participants in this group.

The investigators agree that these protocol deviations will lead to data from these 4 participants to be compromised and hence it will not be analyzed in the final analyses.

ELIGIBILITY:
Inclusion criteria

1. Patients will be 60-85 years of age presenting with major depressive disorder, single or recurrent, as diagnosed by a Mini Neuropsychiatric Interview (MINI) [41].
2. A 17-item Hamilton Depression Rating Scale score of 10-22[42].
3. Participants will be willing and able to attend all 4 training sessions of SSM/HEP, as well as 75% of follow-up sessions.
4. Have sufficient hearing to follow verbal instructions;
5. Have adequate understanding of English in London and English and/or French in Montreal.
6. Able to sit for 45 minutes without discomfort.
7. Willing to remain on the same antidepressants including dosage for the first 12 weeks of the study.

Exclusion criteria

1. Inability to independently provide informed consent.
2. Clinical evidence of dementia as defined by Mini-Cog < 3.a lifetime diagnosis of other mental disorders, including bipolar I or II disorder, primary psychotic disorder (schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder).
3. Substance abuse or dependence within the past 3 months; high risk of suicide (e.g., active suicidal ideation and/or current/recent intent or plan) as assessed by the MINI.
4. Severe personality disorder, that will interfere with their ability to function in a group setting.
5. Substance use disorder as assessed by the MINI.
6. Clinically significant sensory impairment.
7. IQ estimated to be below 70 on the Test of Premorbid Functioning
8. Acutely unstable medical illnesses, including delirium or acute cerebrovascular or cardiovascular events within the last 6 months; having a terminal medical diagnosis with prognosis of less than 12 months.
9. Currently practicing any form of body-mind intervention on a regular basis.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2022-04-09 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms: Hamilton Depression Scale (HAM-D17) | Change from week 0 to week 12 and change from week 0 to week 26.
  The HAM-D17 is a measure of depressive symptoms. Higher scores on this scale indicate greater depression severity; whereas lower scores indicate minimal/no presence of depression. Change in participant scores on this scale throughout the study will be assessed.

SECONDARY OUTCOMES:
Delis-Kaplan Executive Function System (D-KEFS): Verbal Fluency Test | 0 weeks (baseline); 12 weeks; and 26 weeks
  The Verbal Fluency Test of the D-KEFS asks participants to provide responses according to rules set out by 3 sub-tests (letter fluency, category fluency, and category switching). Correct and incorrect responses are scored. The higher number of correct responses and the lower number of incorrect responses is indicative of stronger verbal fluency. A higher number of incorrect responses and/or lower number of correct responses in one of the sub-tests may indicate neurological dysfunction in a corresponding brain region. No global score is generated.
California Verbal Learning Test-II (CVLT-II), Short Form | 0 weeks (baseline); 12 weeks; and 26 weeks
  The CVLT-II is a tool used to assess verbal learning and memory. Scores are determined by recording correct and incorrect responses on each task. Raw scores are used to assess overall performance on the CVLT-II, with higher correct responses and lower incorrect responses indicating good executive functioning.
Rey-Osterrieth Complex Figure-Copy Trial | 0 weeks (baseline); 12 weeks; and 26 weeks
  This neuropsychological test asks participants to draw an image they have been shown after no delay (copying it), a short delay, and a longer delay. The accuracy of each drawn image to the original at each time point is indicative of neurological systems' functioning level.

OTHER OUTCOMES:
Generalized Anxiety Disorder 7-item (GAD-7) scale | 0 weeks (at screening or at baseline); 12 weeks; and 26 weeks
  A measure of anxiety with 7 items scored from 0-3. Higher scores indicate greater depressive symptoms (5-9, mild anxiety; 10-14, moderate anxiety; 15-21 severe anxiety).
Clinical Global Impression (CGI) scale | 0 weeks (baseline); 12 weeks; and 26 weeks
  The CGI is a 3-item scale, psychiatric tool meant to provide an overall picture of a participant's illness severity (1-normal to 7-amongst the most severely ill patients), improvement/change (1-very much improved to 7-very much worse), and therapeutic response (0-marked improvement with no side-effects to 4-unchanged or worse and side-effects outweigh the therapeutic effects). No global score is generated.
Athens Insomnia Scale | 0 weeks (baseline); 12 weeks; and 26 weeks
  The Athens Insomnia Scale is a measure of sleep difficulties with each item representing a different aspect of sleep (e.g. "Overall Quality of Sleep"). Ratings are from 0 to 4, with 0 being no difficulty with the item and 4 being the most difficulty with the item. Higher overall scores on this scale indicate higher difficulties with sleep.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | 0 weeks (baseline); 12 weeks; and 26 weeks
  The WHODAS 2.0 is a 36-item questionnaire assessing a participant's difficulties, due to physical- or mental-health issues, in various activities (e.g. "Self-care") over the past 30 days. Participants provide responses from 1 to 5, with 1 being "None" and 5 being "Extreme or cannot do". Item raw scores, raw domain scores, and domain average scores (out of 5) are generated as well as a "General Disability Score (Total)" and a global average score (out of 5). Higher scores indicate greater difficulty with the item, the domain, overall, or on average.
Euroqol 5 Dimension 5 Level (EQ-5D-5L) | 0 weeks (baseline); 12 weeks; and 26 weeks
  The EQ-5D-5L is a 2 page assessment of a participant's self-rated health state on that day. The first page asks participants to indicate how much difficulty they have in a health dimension (e.g. "Mobility") using one of 5 levels: no problems, slight problems, moderate problems, severe problems, or extreme problems. Higher scores indicate greater severity of problems with a health dimension or overall. The second page asks participants to rate their current health state on a scale from 0 ("the worst health you can imagine") to 100 ("the best health you can imagine"). This section serves as a subjective measure of a participant's own health.
Toronto Side Effects Scale (TSES) | 0 weeks (baseline); 12 weeks; and 26 weeks
  This 32-item scale asks about a broad variety of participant reported side effects. The scale assesses the frequency and intensity of side effects on a 5-point Likert scale, with higher scores indicating greater frequency/severity of the side effect.
Montreal Cognitive Assessment (MoCA; London only) | 0 weeks (baseline); 12 weeks; and 26 weeks
  The MoCA is a brief 30-item measure of different cognitive abilities (e.g. visuospatial ability, short-term memory). Scores range from 0-30, with scores above 26 indicating normal cognitive functioning.
Wechsler Adult Intelligence Scale (WAIS-IV) -Test of premorbid functioning | 0 weeks (baseline); 12 weeks; and 26 weeks
  WAIS-IV-Test of premorbid functioning is a test that assesses cognitive and memory functioning. Performance on this test will be used to estimate a participant's Intelligence Quotient.
Wechsler Adult Intelligence Scale (WAIS-IV)-Digit Span | 0 weeks (baseline); 12 weeks; and 26 weeks
  WAIS-IV-Digit Span is an attention span task involving repeating digits in forward order, backward order, as well as sequencing digits in mind.
Delis-Kaplan Executive Function System (D-KEFS) Color Word Test Conditions 1-3 | 0 weeks (baseline); 12 weeks; and 26 weeks
  D-KEFS Color Word Test is a test of the ability to rapidly name colour patches, rapidly read colour names, and inhibit a response in favor of another response (inhibition trial).
Phenomenology of Consciousness Inventory (PCI) | 12 weeks; and 26 weeks
  The PCI is a self-report measure containing 53 items about an immediately preceding subjective experience, scored on 7-point scales between opposing statements. The items are organized into 21 scales that include altered states of awareness, self-awareness, altered experiences, volitional control, rationality, internal dialogue, positive affect (which includes joy, love and sexual excitement), negative affect (which includes anger, sadness and fear), imagery, attention, memory and arousal. Scores on the scales will be used to assess the degree to which a person has experienced an altered state of consciousness.
Ryff Scales of Psychological Well-Being (SPWB) | 0 weeks (baseline); 12 weeks; and 26 weeks
  SPWB is a self-report measure with 54 short questions that creates scores for six dimensions of psychological well-being: self-acceptance, the establishment of quality ties to others, a sense of autonomy, the pursuit of meaningful goals and a sense of purpose in life, and continued growth and development as a person. This measure is scored on a 6-point scale from "Strongly Disagree" to "Strongly Agree." These scales are regarded as separate dimensions of psychological well-being but can also be aggregated for a global score.
Five Facet Mindfulness Questionnaire (FFMQ) | 0 weeks (baseline); 12 weeks; and 26 weeks
  The FFMQ is a 29-item questionnaire that examines five factors of mindfulness including observe, describe, act with awareness, nonjudge and nonreact. Each question is scored from 1 (never of rarely true) to 5 (very often or always true).
Height | 0 weeks (baseline)
  Participants' heights will be recorded in centimeters.
Weight | 0 weeks (baseline); 12 weeks; and 26 weeks
  Participants' weights will be recorded in kilograms.
Hip and waist circumference | 0 weeks (baseline); 12 weeks; and 26 weeks
  Participants' hip and waist circumferences will be recorded in centimeters.
Medications | 0 weeks (baseline); 12 weeks; and 26 weeks
  Physiological measurement. Will record participants' current list of medication, doses, and how long they have been prescribed/taking the medication.
Blood draw | 0 weeks (baseline) and 12 weeks
  Blood will be taken from participants to measure inflammatory markers, that have been linked to depression, in blood serum.
functional Magnetic Resonance Imaging (fMRI)/Magnetic Resonance Imaging (MRI)/ structural Magnetic Resonance Imaging (sMRI) | 0 weeks (baseline) and 12 weeks
  Physiological measurement. Brain scans will measure neural connectivity and cortical thickness.
Gait (London only) | 0 weeks (baseline); 12 weeks; and 26 weeks
  Outcomes include mean stride length and mean gait velocity. Both stride length and gait speed will be measured using a GAITRite® portable walkway with embedded pressure sensors.
Fall Efficacy Scale - International (FES-I) | 0 weeks (baseline); 12 weeks; and 26 weeks
  The FES-I is a 16-item scale used to assess fear of falling. Scores range from 16-64, with higher scores indicating greater fear of falling.
Mini-Cog | 0 weeks (screening)
  The Mini-Cog is a tool designed for older adults that screens for cognitive impairments. It has two components: 3-item recall and clock drawing. Points are given for correctly recalling items and correctly drawing a clock (e.g. numbers 1-12 present and in clockwise order). Scores range from 0-5, with higher scores indicating normal cognitive functioning, and scores below 3 indicating increased likelihood of dementia.
Patient Health Questionnaire (PHQ-9) | 0 weeks (screening), week 12, and week 26.
  A measure of depression. Scores of: 0-4, no depression; 5-9, mild depression; 10-14, moderate depression; 15-19, moderately severe depression; 20-27, severe depression.
Antidepressant Treatment History Form (ATHF) | 0 weeks (screening)
  The ATHF is a clinical tool used to record and assess the effectiveness of a participant's past treatment(s) for depression (e.g. drug, dose, duration, etc.). In this study, 2 or more rounds of failed or ineffective treatments qualifies the patient as treatment-resistant.
Mini International Neuropsychiatric | 0 weeks (screening)
  A short diagnostic inventory designed to test for assess the presence of 17 common mental health disorders (e.g. Major Depressive Disorder, Manic Episode, or Alcohol Use Disorder).
Cumulative Illness Rating Scale - Geriatrics (CIRS-G) | 0 weeks (baseline)
  An assessment for 14 body systems. Each are rated on a scale of 0-4; with 0 representing no issue to 4 representing sever problems with that system. A higher score, overall, indicates greater problems or greater severity of problems with the various health systems.
Time Trade Off (TTO) | Weeks 0, week 12, week 24.
  An assessor of the quality of the participants health rated from 0 to 10. Lower numbers indicate a poorer state of health while higher numbers indicate a better state of health.
Index of Vascular Burden | 0 weeks (baseline)
  An assessment of obesity, hypertension, smoking and diabetes. Each item is scored as 0 for no or 1 for yes and a total score is calculated ranging from 0 to 4.
Socioeconomic Status Index (SES) | 0 weeks (baseline)
  An assessment of SES that includes annual household income from the previous year, number of individuals in household and personal income in the previous year.
Acti watch | Weeks -2 and 14.
  In Montreal only the GENEActiv Original wrist actigraphy device will record rest-activity rhythm.
Likert Scale | Week 12
  An assessment of how participants enjoyed the intervention rated from 0 to 10. Participants are requested to indicate if they strongly disagree, disagree, neutral, agree, or strongly agree to statements about the programs helpfulness, convenience, instructors, how enjoyable the program was and if they now feel happier compared to before the intervention.
Qualitative Side Effects | Weeks 12 and 26.
  Participants are asked to describe any adverse events they experienced while participating in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data with researchers who are not currently involved with the project. The Co-PIs, Co-Is, and research staff at Western and McGill sites will have access to all participant data through the secure online system, REDCap.

REFERENCES:
- [Derived] Peckham SB, Ionson E, Nassim M, Ojha K, Palaniyappan L, Gati J, Theberge J, Lazosky A, Speechley M, Baruss I, Rej S, Vasudev A. Sahaj Samadhi meditation vs a Health Enhancement Program in improving late-life depression severity and executive function: study protocol for a two-site, randomized controlled trial. Trials. 2019 Oct 24;20(1):605. doi: 10.1186/s13063-019-3682-z. PMID 31651355